CLINICAL TRIAL: NCT03771404
Title: Evaluation of Non-small Cell Lung Carcinoma Genetic Heterogeneity in Patients With Operable Early Stage Disease and Prediction of Clinical Relapse Using a Personalized "Liquid Biopsy"
Brief Title: NSCLC Heterogeneity in Early Stage Patients and Prediction of Relapse Using a Personalized "Liquid Biopsy"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CT/17.01
Record Dates: First submitted 2018-11-14; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; Tumor heterogeneity; liquid biopsy; CTCs; ctDNA; NGS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Operable (stages I-IIIA) NSCLC (Other): For Operable (stages I-IIIA) NSCLC Patients, blood sampling and tissue samples of the primary tumor as well as the regional involved lymph nodes and, in selected patients, from biopsies from metastasis
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — Patients' peripheral blood will be obtained before the surgical excision of the primary tumor as well as 1-month post-op and every 3-6 months thereafter until disease progression and upon disease relapse for the evaluation of ctDNA and CTCs. Different sites of the primary tumor as well as the regional involved lymph nodes and, in selected patients, biopsies from metastatic sites will be genotyped by NGS as well.
  Other Names: primary tumor sampling after surgery; biopsy from metastatic sites in selected patetients

SUMMARY:
The purpose of his study is to investigate the intra tumor heterogeneity of the primary tumor and the involved lymph nodes from patients with resectable NSCLC, to detect primary tumor genetic alternations using "liquid biopsy" during the patients' clinical follow up and to correlate the "liquid biopsy" information with the disease recurrence.

DETAILED DESCRIPTION:
Lung cancer is the most common cancer in the world. In operable early stage patients NSCLS can be curable, but even after complete primary tumor resection, about 45% of early stage patients develop local or distant recurrence within 8-18 months. Recent studies have established that targeted therapies may fail to cure the disease because of tumor heterogeneity. The presence of genetic heterogeneity in different portions of a tumor have demonstrated its importance in tumor biology suggesting that pre-existing genetically different sub clones may be selected by therapy or differentially involved in the metastatic process, leading to treatment failure.

The relationship of tumor heterogeneity with the poor clinical outcome suggests that its assessment could provide interesting and useful clinical information, especially, in terms of prognosis and treatment selection. It is now, well established that during the evolution of tumor new cellular clones could be emerged which differ genetically from the molecular signature of tumor cells evaluated at the time of initial diagnosis. This molecular evolution may further contribute to the tumor heterogeneity during the disease progression. The evaluation of the real-time molecular tumor heterogeneity requires repeated re-biopsies during the different clinical phases of NSCLC which, however, are invasive and not, always, feasible. This problem can be by-passed by the use of tumor-originating elements in the plasma and among these cellular products the isolation and analysis of cell tumor DNA (ctDNA) and the characterization of Circulating Tumor Cells (CTCs) represent important tools for identification and monitoring of molecular tumor alterations in cancer patients, representing what the investigators call "liquid biopsy". ctDNA is originated from cellular necrosis due to increased tumoral cellular turnover and cellular ischemia as well as from apoptosis of tumor cells or lysis of Circulating Tumor Cells (CTCs). On the other hand, the CTCs, which designate the cells circulating in the blood, can be detected in several tumor types, irrespectively of the clinical phase, and their detection has been correlated with disease progression and treatment resistance. Therefore, the concomitant analysis of both ctDNA and CTCs could permit to better evaluate the genetic heterogeneity of the tumor since they continuously released from tumor cells throughout the clinical course of the disease and is considered to be proportional to tumor burden and tumor progression at each time-point.

This is a multicenter, single arm, non-randomized translational research study. Patients with operable NSCLC will be enrolled in the study. Patients' peripheral blood will be obtained before the surgical excision of the primary tumor as well as 1-month post-op and every 3-6 months thereafter until disease progression and upon disease relapse for the evaluation of ctDNA and CTCs. Different sites of the primary tumor as well as the regional involved lymph nodes and, in selected patients, biopsies from metastatic sites will be genotyped by NGS as well.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC (adenocarcinoma and squamous cell carcinoma).
* Age ≥ 18 years
* Operable (stages I-IIIA) NSCLC
* Patients with signed written informed consent obtained according to local guidelines

Exclusion Criteria:

* Patients < 18 years
* Patients with non operable NSCLC (regardless of disease stage)
* Patients who have any current or prior medical condition that may interfere with the conduct of the study or the evaluation of its results in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate whether the individual patient's molecular landscape of ctDNA and CTCs could be reliable biomarkers for the early prediction of disease relapse. | Up to 2 years
  The initial tumor of all patients will be submitted to Next Generation Sequencing (NGS) in order to detect mutations and copy-number variations to the following set of genes: AKT1, KRAS, NRAS, BRAF, DDR2, EGFR, FGFR1, ERBB2 (HER2), MEK1, MET, PIK3CA, PTEN, TP53, MDM2, SOX2 and P63. Detected mutations will be monitored longitudinally in ctDNA from patient's blood samples by ddPCR, for a 2-year period or until PD. For each subject, molecular analysis results will be correlated with its clinical outcome in terms of time to disease progression (PFS). CTCs will be isolated based on the cell's size. CTCs isolated by ISET will be phenotypically characterized to define their proliferative, apoptotic, EMT status as well as their immune profile using antibodies and immunofluorescent staining. CTCs isolated by PARSORTIX will be analyzed for the detection of specific genetic changes present in the primary tumor (see NGS analysis of primary tumor) using either qRT-PCR or FISH analysis.

SECONDARY OUTCOMES:
To investigate the genetic heterogeneity in resectable NSCLC | Up to 2 years
  The initial tumor of all patients will be submitted to Next Generation Sequencing (NGS) in order to detect mutations and copy-number variations to the following set of genes: AKT1, KRAS, NRAS, BRAF, DDR2, EGFR, FGFR1, ERBB2 (HER2), MEK1, MET, PIK3CA, PTEN, TP53, MDM2, SOX2 and P63.
To monitor using "liquid biopsy" the tumor clonal evolution during the post operation period and define a correlation between the genotype of the primary tumor and the emergence of molecularly different clones | Up to 2 years
  The initial tumor of all patients will be submitted to Next Generation Sequencing (NGS) in order to detect mutations and copy-number variations to the following set of genes: AKT1, KRAS, NRAS, BRAF, DDR2, EGFR, FGFR1, ERBB2 (HER2), MEK1, MET, PIK3CA, PTEN, TP53, MDM2, SOX2 and P63. Detected mutations will be monitored longitudinally in ctDNA from patient's blood samples by droplet digital Polymerase Chain Reaction (ddPCR), for a 2-year period or until PD.
To investigate the potential of longitudinal "liquid biopsy" to predict the genetic profile of metastasis | Up to 2 years
  The initial tumor of all patients will be submitted to Next Generation Sequencing (NGS) in order to detect mutations and copy-number variations to the following set of genes: AKT1, KRAS, NRAS, BRAF, DDR2, EGFR, FGFR1, ERBB2 (HER2), MEK1, MET, PIK3CA, PTEN, TP53, MDM2, SOX2 and P63. Detected mutations will be monitored longitudinally in ctDNA from patient's blood samples by droplet digital Polymerase Chain Reaction (ddPCR), for a 2-year period or until PD. Moreover, in patients where metastasis re-biopsy is feasible the metastasis tumor will be submitted to Next Generation Sequencing (NGS) in order to detect mutations and copy-number variations to the set of genes mentioned above. Correlation between the molecular analysis of the primary tumor, the ctDNA and the metastasis tumor will reveal whether longitudinal liquid biopsy can predict the metastasis genetic profile.

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Kotsakis, MD, PhD, Principal Investigator — Chairman of the Lung Cancer Working Group of the HORG
Locations (6):
- Greece (6):
  - 2nd Pneumological Dept, GNA "Sotiria", Athens, Attica
  - 7th Pneumological Dept, GNA "Sotiria", Athens, Attica
  - Thoracic Surgery Dept, GNA "Sotiria", Athens, Attica
  - Thoracic Surgery Clinic, "Hygeia" Hospital, Athens, Attica
  - Oncology Unit, 3rd Department of Medicine Athens University School of Medicine Athens, GNA "Sotiria", Athens
  - IASO General Hospital, Athens

IPD SHARING:
Plan to Share IPD: No